CLINICAL TRIAL: NCT04231383
Title: Evaluation of the Relationship Between Dental Caries-related Pain and Inflammation and Growth Parameters in Preschool Children
Brief Title: Evaluation of the Relationship Between Dental Caries and Growth Parameters in Preschool Children
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Basak Gunay, research asistant, Bezmialem Vakif University
Other Study IDs: 8.2019/7
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Dental Caries in Children
Keywords: Dental caries; IGF-1; IGFBP-3; anthropometry; sleeping
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: dental caries, growth parametres — The comparison of growth parameters before and after 6 months of treatment of dental caries will be compared.
  Children's Sleep Habits Questionnaire and Early Childhood Oral Health Impact Scale will be compared before and at the 6th month of dental treatment.

SUMMARY:
Untreated dental caries are very common in preschool children. Pain and inflammation due to dental caries have been reported to affect eating and sleeping disorders, affecting growth and development. The aim of this study was to compare the changes in serum IGF-1 and IGFBP-3 levels, height and weight gain before and after treatment in patients with dental caries-related inflammation and pain in preschool children and to compare these children with children without dental caries. Thirty children aged between 3-6 years with dental caries with pulp were identified using ICDAS II and dmft index as the study group.30 children dental caries including pulp, will be included using the same indices as the control group. In the study group, serum IGF-1 and IGFBP-3 levels and anthropometric measurements will be determined before and at the 6th month after treatment. In the control group, serum IGF-1 and IGFBP-3 levels and anthropometric measurements will be determined at the 6th month following the first dental examination. IGF-1, IGFBP-3 and anthropometric measurements will be compared between first dental examination and 6th month values in the study and control groups, and between first dental examination and 6th month time points between the groups.

DETAILED DESCRIPTION:
In addition to growth parameters, the Children's Sleeping Habits Questionnaire and the Early Childhood Oral Health Impact Scale will be compared before the 6th month of dental treatment and compared

ELIGIBILITY:
Inclusion Criteria:

For study group

1. (3-6 years) preschool children
2. Children whose dental treatments are indicated under general anesthesia
3. Children with primary dentition
4. Children with early childhood caries (dmft index d≥ 3)
5. Children with symptoms of pulpitis or periapical infection in at least one tooth
6. Children with dental problems at least in the last 6 months
7. Volunteering to participate in the study. For the control group,

1- (3-6 years) preschool children 2-Children with primary dentition 3- Children without pulpitis symptoms or periapical infection during dental examination 4-Volunteering to participate in the study.

Exclusion Criteria:

1. Children who do not show adequate compliance during blood sampling
2. Consent form is not signed
3. Children with chronic and systemic diseases that may affect growth and development
4. Children using anti-inflammatory
5. Patients with physical and mental disabilities
6. Patients using corticosteroids in the last 6 months
7. If a child is diagnosed with any of the these diseases during the study

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Thirty children aged between 3-6 years with dental caries with pulp were identified using ICDAS II and dmft index as the study group.30 children dental caries including pulp, will be included using the same indices as the control group
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-04-15 (Estimated); Study Completion 2020-06-15 (Estimated)

PRIMARY OUTCOMES:
Growth parameters | before dental treatment
  In the study group, serum IGF-1 and IGFBP-3 levels and anthropometric measurements will be determined before and at the 6th month after treatment. In the control group, serum IGF-1 and IGFBP-3 levels and anthropometric measurements will be determined at the 6th month following the first dental examination. IGF-1, IGFBP-3 and anthropometric measurements will be compared between first dental examination and 6th month values in the study and control groups, and between first dental examination and 6th month time points between the groups.
Growth parameters | 6 months after dental treatment
  In the study group, serum IGF-1 and IGFBP-3 levels and anthropometric measurements will be determined before and at the 6th month after treatment. In the control group, serum IGF-1 and IGFBP-3 levels and anthropometric measurements will be determined at the 6th month following the first dental examination. IGF-1, IGFBP-3 and anthropometric measurements will be compared between first dental examination and 6th month values in the study and control groups, and between first dental examination and 6th month time points between the groups.

SECONDARY OUTCOMES:
Children's Sleep Habits Questionnaire | before dental treatment
  In the study group Children's Sleep Habits Questionnaire will be compared before, after the a week and 6th month of dental treatment.In the control group Children's Sleep Habits Questionnaire will be compared before, after the a week and 6th month of dental treatment
Children's Sleep Habits Questionnaire | a week after dental treatment
  In the study group Children's Sleep Habits Questionnaire will be compared before, after the a week and 6th month of dental treatment.In the control group Children's Sleep Habits Questionnaire will be compared before, after the a week and 6th month of dental treatment
Children's Sleep Habits Questionnaire | 6 months after dental treatment
  In the study group Children's Sleep Habits Questionnaire will be compared before, after the a week and 6th month of dental treatment.In the control group Children's Sleep Habits Questionnaire will be compared before, after the a week and 6th month of dental treatment
Early Childhood Oral Health Impact Scale | before dental treatment
  n the study Early Childhood Oral Health Impact Scale will be compared before, after the a week and 6th month of dental treatment.In the control group Early Childhood Oral Health Impact Scale will be compared before, after the a week and 6th month of dental treatment
Early Childhood Oral Health Impact Scale | a week after dental treatment
  n the study Early Childhood Oral Health Impact Scale will be compared before, after the a week and 6th month of dental treatment.In the control group Early Childhood Oral Health Impact Scale will be compared before, after the a week and 6th month of dental treatment
Early Childhood Oral Health Impact Scale | 6 months after dental treatment
  n the study Early Childhood Oral Health Impact Scale will be compared before, after the a week and 6th month of dental treatment.In the control group Early Childhood Oral Health Impact Scale will be compared before, after the a week and 6th month of dental treatment

CONTACTS AND LOCATIONS:
Overall Officials: Basak Gunay, Principal Investigator — Bezmialem Vakif University; Mustafa Sarp Kaya, Study Director — Bezmialem Vakif University; Ilker Tolga Ozgen, Study Chair — Bezmialem Vakif University
Locations (1):
- Basak Gunay, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alkarimi HA, Watt RG, Pikhart H, Jawadi AH, Sheiham A, Tsakos G. Impact of treating dental caries on schoolchildren's anthropometric, dental, satisfaction and appetite outcomes: a randomized controlled trial. BMC Public Health. 2012 Aug 29;12:706. doi: 10.1186/1471-2458-12-706. PMID 22928903
- [Background] Ersoy B, Yuceturk AV, Taneli F, Urk V, Uyanik BS. Changes in growth pattern, body composition and biochemical markers of growth after adenotonsillectomy in prepubertal children. Int J Pediatr Otorhinolaryngol. 2005 Sep;69(9):1175-81. doi: 10.1016/j.ijporl.2005.02.020. PMID 15885810
- [Background] Duijster D, Sheiham A, Hobdell MH, Itchon G, Monse B. Associations between oral health-related impacts and rate of weight gain after extraction of pulpally involved teeth in underweight preschool Filipino children. BMC Public Health. 2013 Jun 3;13:533. doi: 10.1186/1471-2458-13-533. PMID 23731717